CLINICAL TRIAL: NCT05835908
Title: Follow-up of Patients Referred to Unscheduled Care Centers by the Emergency Call Center in the Haut-Rhin Department, France
Acronym: CSNP68
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 1290
Record Dates: First submitted 2023-04-19; First posted 2023-04-28 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2023-10

CONDITIONS: Unscheduled Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient who contacted the Emergency Call Center and were referred to an Unscheduled Care Center
  Interventions: Other: Phone questionnaire

INTERVENTIONS:
Other: Phone questionnaire — Patients will be contacted by the investigator to collect information regarding follow-up from the initial call to the Emergency call center until the patient is taken care of in the health care facility to which he/she has been admitted.

SUMMARY:
The objective of this study is to determine the follow-up of patients who were referred by the Emergency Call Center of the Haut-Rhin department to an Unscheduled Care Centers (UCC) and to determine whether they actuallly went to a UCC following their call, or if they were taken in charge by another care facility.

DETAILED DESCRIPTION:
Conduct of research:

Patients who contacted the emergency call center and were referred to an unscheduled care center in the Haut-Rhin will be contacted by mail in the first instance. Ten to fifteen days after the call to the emergency call center, the investigator will contact the patient by phone, during which he/she will ask for the patient's oral consent to participate in the research and collect follow-up data using a standardized questionnaire.

If the investigator is unable to reach the patient, further attempts will be made to call the patient up to 30 days after the initial call. If there is no response after this time, patients will not be included the study.

ELIGIBILITY:
Inclusion Criteria:

* Call to the Emergency Call Centre of the Haut-Rhin department by an adult (age ≥ 18 years)
* Referral to the Unscheduled Care Center by the Emergency Call Center

Non-inclusion criteria:

* Patient who does not answer phone within 30 days of call to the Emergency Call Center
* Patient who refuses to participate in the study
* Call for someone other than him or herself (except when a parent calls for his or her minor child)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who contacted the Emergency Call Center and were referred to an Unscheduled Care Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-17 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Phone questionnaire | Up to 30 days following the call to the Emergency call center
  Patients will be contacted by the investigator to collect information regarding follow-up from the initial call to the Emergency call center until the patient is taken care of in the health care facility to which he/she has been admitted. Information will be collected on: time and day of the call to the Emergency call center; reason for call; understanding of the instructions given by the call center agent; delay between the call to the Emergency call centre and the visit to the care facility; and, if applicable, the reason why the patient did not go to the UCC.

CONTACTS AND LOCATIONS:
Locations (1):
- GHRMSA, Mulhouse, Haut-Rhin, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study results — https://ecrin.app.unistra.fr/search/notice/view/ecrin-ori-383707